CLINICAL TRIAL: NCT00455923
Title: SERETIDE vs FLIXOTIDE in Mild Persistent Asthma (GINAII)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: SAM103976
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: asthma; exacerbation; persistent; bronchial hyperresponsiveness; mild; GINAII
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity; Lymphoma, Follicular | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seretide (Experimental): Eligible participants received a starting dose of 50/100 mcg Seretide (combination of Sal/FP) via Diskus inhaler, twice daily. During the first 6 months, when the asthma was unstable/uncontrolled, dose was increased in a stepwise fashion to 50/250 mcg and 50/500 mcg (if still unstable). After the initial 6 months, the treatment was fixed without further changes. The total treatment period was 18 months.
  Interventions: Drug: Seretide
- Flixotide (Experimental): Eligible participants received a starting dose of 100 mcg Flixotide (FP only) via Diskus inhaler, twice daily. During the first 6 months, when the asthma was unstable/uncontrolled, dose was increased in a stepwise fashion to 250 mcg and 500 mcg (if still unstable). After the initial 6 months, the treatment was fixed without further changes. The total treatment period was 18 months.
  Interventions: Drug: Flixotide

INTERVENTIONS:
Drug: Seretide — Seretide
  Arms: Seretide
Drug: Flixotide — Flixotide
  Arms: Flixotide

SUMMARY:
An 18 months randomised double-blind study with two parallel arms with start dose of inhaled SERETIDE 50/100mcg BD or FLIXOTIDE 100mcg BD, Phase I is 6 months where the patient will be up-titrated until well controlled is achieved, After 6 months the treatment continues without changes during 9 months = PhaseII. The aim is to investigate and evaluate the assumption that the combination therapy with SERETIDE controls mild persistent asthma better than inhaled corticosteroids(FLIXOTIDE) alone.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give informed consent.
* Males or females aged 18-70.
* Able to understand and complete dairy cards.
* Mild persistent asthma according to GINA. In addition, at randomisation subjects were required to have: 1. Day time symptoms more than once a week but not every day. 2. Night-time symptoms not more than once a week. 3. FEV1 >80% predicted 4. PC20 <8mg/mL

Exclusion Criteria:

* Change to regular asthma medication in 4-weeks prior to visit 1.
* Use of oral, depot or parenteral corticosteroids within 8 weeks of visit 1.
* Lower respiratory tract within 4 weeks of Visit 1
* Received investigational study drug within 4 weeks of visit
* Smoking history of >10 pack years of more.
* Serious uncontrolled disease.
* Medical conditions or medications known to affect the assessments or endpoints.
* Evidence of alcohol or drug abuse.
* Known pregnancy or planned pregnancy.
* Known or suspected hypersensitivity to inhaled corticosteroids, beta-agonists or lactose.
* Previous enrollment in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05-03 (Actual); Primary Completion 2007-07-31 (Actual); Study Completion 2007-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Luleå, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center with two sites in Sweden from May 2005 to July 2007. Seretide Diskus®, Flixotide® and Ventoline Diskus® are the registered products of GlaxoSmithKline.
Groups:
- Seretide: Eligible participants received a starting dose of 50/100 micrograms (mcg) Seretide (combination of salmeterol/fluticasone propionate (Sal/FP) via Diskus inhaler, twice daily. During the first 6 months, when the asthma was unstable/uncontrolled, dose was increased in a stepwise fashion to 50/250 mcg and 50/500 mcg (if still unstable). After the initial 6 months, the treatment was fixed without further changes. The total treatment period was 18 months.
Period: Overall Study
Arm/Group | Seretide | Flixotide
Started | 50 | 50
Completed | 47 | 47
Not Completed | 3 | 3
Not completed — Pregnancy | 0 | 2
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seretide | Flixotide | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants]
  >=18 to 70 years | 50 | 50 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 18 | 19 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Arm With a Need for an Increase in Study Medication
Description: During the first 6 months, when the asthma was unstable/uncontrolled, dose of Seretide (Sal/FP) was increased from 50/100 mcg in a stepwise fashion to 50/250 mcg and 50/500 mcg (if still unstable). Also, dose of Flixotide (FP only), was increased from 100 mcg to 250 mcg and 500 mcg (if still unstable). After the initial 6 months, the treatment was fixed without further changes. The total treatment period was 18 months. Number of participants in each arm with a need for an increase in study medication are presented.
Time Frame: Up to 18 months
Population: Intent-to-Treat (ITT) Population which comprised of all participants who were randomized and received at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Seretide | Flixotide
Number analyzed (Participants) | 50 | 50
Participants | 29 | 29

2. Secondary Outcome: Absolute Bronchial Hyper-responsiveness up to 18 Months
Description: Data for this outcome measure was not collected.
Time Frame: Up to 18 months
Population: Data for this outcome measure was not collected.
Arm/Group | Seretide | Flixotide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Bronchial Hyper-responsiveness From Baseline to 18 Months
Description: Data for this outcome measure was not collected.
Time Frame: Baseline (Day 0) to 18 months
Population: ITT population. Data for this outcome measure was not collected.
Arm/Group | Seretide | Flixotide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Symptom-free Days and Nights Without Use of Rescue Medication
Description: The rescue medications used for exacerbations included Ventoline Diskus® 200 mcg/dose inhalations as required and oral Prednisolone 25 mg per day for five days, and when necessary, ten days. Data for this outcome measure was not collected.
Time Frame: Up to 18 months
Population: ITT population. Data for this outcome measure was not collected.
Arm/Group | Seretide | Flixotide
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Exacerbations: in Total and by Degree of Severity
Description: Severe exacerbation: needed hospitalization/emergency unit visit. Moderate exacerbation: Needed oral cortico-steroid or adding inhaled Flixotide to maintenance study medicine; decrease in morning or evening peak expiratory flow (PEF) > 30% during ≥ 2 following days from Baseline (Day 0). Mild exacerbation: any night symptoms ≥ 3 consecutive, or night symptoms ≥ 2 consecutive nights in case symptoms have been scored ≥ 2 during at least one night, Day symptoms scored ≥ 2 during ≥ 4 following days, or Day symptoms scored ≥ 3 during ≥ 3 following days, or Day symptoms scored ≥ 4 during ≥ 2 following days, or rescue medication use ≥ 2 occasions per day for ≥ 4 following days, or rescue medication use ≥ 3 occasions per day for ≥ 3 following days, or rescue medication use ≥ 4 occasions per day for ≥ 2 following days, or decrease in morning/evening PEF >20% during ≥ 2 following days from Baseline (Day 0). Number of total exacerbations and severe, moderate and mild exacerbations are presented.
Time Frame: Up to 18 months
Population: ITT Population.
Measure: Number; unit: Exacerbations
Arm/Group | Seretide | Flixotide
Number analyzed (Participants) | 50 | 50
Exacerbations
  Total exacerbations | 42 | 74
  Severe exacerbations | 0 | 1
  Moderate exacerbations | 12 | 21
  Mild exacerbations | 30 | 52

6. Secondary Outcome: Time to Increase of Study Medication
Description: Data for this outcome measure was not collected.
Time Frame: Up to 6 months
Population: ITT population. Data for this outcome measure was not collected.
Arm/Group | Seretide | Flixotide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: Adverse events (Serious adverse events and non-serious adverse events) were collected and are reported for the ITT Population.
Arm/Group | Seretide | Flixotide
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/50
Other Adverse Events (participants affected / at risk) | 48/50 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seretide (N=50) | Flixotide (N=50)
Colon diverticulitis (Gastrointestinal disorders) | 1 | 0
Migraine/headache (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seretide (N=50) | Flixotide (N=50)
Common cold (Infections and infestations) | 45 | 39
Upper airway infections (Infections and infestations) | 14 | 15
Headache (Nervous system disorders) | 8 | 7
Gastroenteritis (Infections and infestations) | 9 | 8
Pharyngitis (Infections and infestations) | 7 | 4
Bronchitis (Infections and infestations) | 4 | 5
Mouth candida (Infections and infestations) | 2 | 4
Sinusitis (Infections and infestations) | 3 | 1
Upper back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Chest pain (General disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.